CLINICAL TRIAL: NCT03276988
Title: A Prospective, Open-label, Dose Escalation,(Phase 1); Prospective, Randomized, Evaluator Blinded, Active-controlled, 2-sequence, 2-period, 2-treatment, Crossover(Phase 2); Phase 1/2 Clinical Trial to Evaluate the Tolerability, Pharmacokinetics, Safety and Efficacy of GX-30 Administered Intramuscularly in Patients Underwent Total Thyroidectomy or Near Total Thyroidectomy
Brief Title: Tolerability, Safety and Pharmacokinetics Study of GX-30 in Total Thyroidectomy or Near Total Thyroidectomy Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Collaborators: Symyoo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: GX30_P1/2
Record Dates: First submitted 2017-09-04; First posted 2017-09-08 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Total Thyroidectomy; Near-total Thyroidectomy
Keywords: Thyroid cancer; Thyroidectomy; rhTSH; GX-30
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Thyrotropin Alfa

STUDY DESIGN:
Intervention Model Description: The Part A (Phase 1) of study has been completed in which 3 single or multiple sequentially assenting doses of GX-30 were investigated. The Part B (Phase 2) is recruiting in current in which each study participant will receive the same multiple doses of GX-30 and THYROGEN® but at different period.
Who Masked: Participant, Outcomes Assessor
Masking Description: At Part B, Both independent central efficacy assessors and participants will be masked. Investigators will be unmasked. (The Part A was open-label.)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part B - Sequence A (Other): Period 1 GX-30 0.9mg x 2 (Day 1 and Day 2), IM injection. Period 2 THYROGEN® 0.9mg x 2 (Day 1 and Day 2), IM injection
  Interventions: Drug: Period 1 GX-30, Period 2 THYROGEN®
- Part B - Sequence B (Other): Period 1 THYROGEN® 0.9mg x 2 (Day 1 and Day 2), IM injection. Period 2 GX-30 0.9mg x 2 (Day 1 and Day 2), IM injection
  Interventions: Drug: Period 1 THYROGEN®, Period 2 GX-30

INTERVENTIONS:
Drug: Period 1 GX-30, Period 2 THYROGEN® — Part B - Sequence A. GX-30 0.9mg will be administered at Day 1 and Day 2 in Period 1. After wash-out period of 2 to 3 weeks, THYROGEN® 0.9mg will be administered in Period 2.
  Other Names: Thyrotropin alpha
  Arms: Part B - Sequence A
Drug: Period 1 THYROGEN®, Period 2 GX-30 — Part B - Sequence B. THYROGEN® 0.9mg will be administered at Day 1 and Day 2 in Period 1. After wash-out period of 2 to 3 weeks, GX-30 0.9mg will be administered in Period 2.
  Other Names: Thyrotropin alpha
  Arms: Part B - Sequence B

SUMMARY:
This study is designed as a combination of phase 1 (Part A) and phase 2 (Part B). The purpose of Part A was to determine the safety, tolerability, and pharmacokinetics in patients with total thyroidectomy or near total thyroidectomy of GX-30 and it has been completed. The Part B is currently recruiting and will investigate the efficacy and safety of GX-30 compared with THYROGEN®.

DETAILED DESCRIPTION:
Recombinant human TSH was developed to provide TSH stimulation without withdrawal of thyroid hormone. Radioiodine ablation and diagnosis with rhTSH became the standard of care treatment for patients with differentiated thyroid cancer. Stably supplying rhTSH has been the unmet need for management and follow-up procedure for thyroid remnant. GX-30 is an investigational product, developed to provide inexpensive rhTSH to patients in order to ensure stable supply of rhTSH.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who voluntarily consented, after listing enough explanation for this study and investigational product.
* Minimum 19 years old.
* Minimum 50kg of body weight.
* Patients who had undergone total thyroidectomy or near total thyroidectomy due to differentiated thyroid carcinoma.
* Patient undergoing thyroid hormone administration.

Exclusion Criteria:

* Thyroid cancer excluding differentiated thyroid carcinoma.
* Thyroidectomy excluding total thyroidectomy and near total thyroidectomy.
* Patients with heart, renal, or liver failure.
* Patients with ischemic stroke or the history of ischemic stroke.
* Smoker or Ex-smoker with less than 3 months of stopping
* Patients with migraine or the history of migraine.
* Patients that the researchers do not think fit into the group, including patients failed in compliance assessment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant or lactating women will be excluded. Women of childbearing potential who agreed to use a medically appropriate conceptional method till 6 months after study completion may be enrolled.
Enrollment: 8 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Efficacy (Part B) | at each Day 4, period 1 and period 2.
  I-123 Whole body scan image classification

SECONDARY OUTCOMES:
TSH concentration (Part B) | Baseline, Day 1 to Day 8.
  TSH concentration for Pharmacokinetics assessment
ADA (Part B) | Baseline, Day 1 and 15 of Period 2
  Anti-Drug Antibody detection
Tg concentration (Part B) | Baseline, Day 1 to Day 5
  Thyroglobulin concentration for secondary efficacy assessment
T3, free T4 concentration (Part B) | Baseline, Day 1, 2, 5 of each period and Day 15 of period 2.
  Thyroid hormones concentration for pharmacodynamic assessment
Adverse events (Part B) | through study completion, average of 6 weeks.
  Safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: Mu Il Kang, M.D., Ph. D., Principal Investigator — Seoul St. Mary's Hospital
Locations (5):
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Korea University Anam Hospital, Seoul
  - Seoul Asan Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goel R, Raju R, Maharudraiah J, Sameer Kumar GS, Ghosh K, Kumar A, Lakshmi TP, Sharma J, Sharma R, Balakrishnan L, Pan A, Kandasamy K, Christopher R, Krishna V, Mohan SS, Harsha HC, Mathur PP, Pandey A, Keshava Prasad TS. A Signaling Network of Thyroid-Stimulating Hormone. J Proteomics Bioinform. 2011 Oct 29;4:10.4172/jpb.1000195. doi: 10.4172/jpb.1000195. PMID 24255551
- [Background] Meier CA, Braverman LE, Ebner SA, Veronikis I, Daniels GH, Ross DS, Deraska DJ, Davies TF, Valentine M, DeGroot LJ, et al. Diagnostic use of recombinant human thyrotropin in patients with thyroid carcinoma (phase I/II study). J Clin Endocrinol Metab. 1994 Jan;78(1):188-96. doi: 10.1210/jcem.78.1.8288703.
- [Background] Torres MS, Ramirez L, Simkin PH, Braverman LE, Emerson CH. Effect of various doses of recombinant human thyrotropin on the thyroid radioactive iodine uptake and serum levels of thyroid hormones and thyroglobulin in normal subjects. J Clin Endocrinol Metab. 2001 Apr;86(4):1660-4. doi: 10.1210/jcem.86.4.7405. PMID 11297600
- [Background] Ladenson PW, Braverman LE, Mazzaferri EL, Brucker-Davis F, Cooper DS, Garber JR, Wondisford FE, Davies TF, DeGroot LJ, Daniels GH, Ross DS, Weintraub BD. Comparison of administration of recombinant human thyrotropin with withdrawal of thyroid hormone for radioactive iodine scanning in patients with thyroid carcinoma. N Engl J Med. 1997 Sep 25;337(13):888-96. doi: 10.1056/NEJM199709253371304. PMID 9302303
- [Background] Haugen BR, Pacini F, Reiners C, Schlumberger M, Ladenson PW, Sherman SI, Cooper DS, Graham KE, Braverman LE, Skarulis MC, Davies TF, DeGroot LJ, Mazzaferri EL, Daniels GH, Ross DS, Luster M, Samuels MH, Becker DV, Maxon HR 3rd, Cavalieri RR, Spencer CA, McEllin K, Weintraub BD, Ridgway EC. A comparison of recombinant human thyrotropin and thyroid hormone withdrawal for the detection of thyroid remnant or cancer. J Clin Endocrinol Metab. 1999 Nov;84(11):3877-85. doi: 10.1210/jcem.84.11.6094. PMID 10566623
- See also: Park DJ. Thyroid and Hydrogen Peroxide. Hanyang Med Rev 2012;32:187-91 — https://synapse.koreamed.org/DOIx.php?id=10.7599/hmr.2012.32.4.187